CLINICAL TRIAL: NCT00920153
Title: Study Characterizing the Impact of Different Therapeutic Strategies on Event Occurrence at 2 Years, 5 Years, 10 Years, and 15 Years, According to Prognostic Groups in Patients With Hodgkin Lymphoma
Brief Title: Three Different Therapy Regimens in Treating Patients With Previously Untreated Hodgkin Lymphoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Other new drugs
Sponsor: French Innovative Leukemia Organisation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LH 2007
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-07

CONDITIONS: Lymphoma
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Bleomycin; ABVD protocol; Carmustine; Cisplatin; Cytarabine; Dacarbazine; Dexamethasone; Doxorubicin; Etoposide; Gemcitabine; Ifosfamide; Melphalan; Methylprednisolone; Mitoguazone; Vincristine; Vindesine; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (favorable prognosis) (Experimental): Patients receive ABVD and VABEM chemotherapy.
  Interventions: Biological: bleomycin sulfate; Drug: ABVD regimen; Drug: carmustine; Drug: dacarbazine; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: methylprednisolone; Drug: vincristine sulfate; Drug: vindesine
- Group 2 (intermediate prognosis) (Experimental): Patients receive ABVD and VABEM chemotherapy.
  Interventions: Biological: bleomycin sulfate; Drug: ABVD regimen; Drug: carmustine; Drug: dacarbazine; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: methylprednisolone; Drug: vincristine sulfate; Drug: vindesine
- Group 3 (poor prognosis) (Experimental): Patients receive VABEM, CEO, BEAM, and MINE chemotherapy. Patients also undergo allogeneic or autologous stem cell transplantation.
  Interventions: Drug: carmustine; Drug: cisplatin; Drug: cytarabine; Drug: dexamethasone; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: gemcitabine hydrochloride; Drug: ifosfamide; Drug: melphalan; Drug: methylprednisolone; Drug: mitoguazone; Drug: vindesine; Drug: vinorelbine tartrate; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: autologous hematopoietic stem cell transplantation

INTERVENTIONS:
Biological: bleomycin sulfate — Given IV
  Arms: Group 1 (favorable prognosis); Group 2 (intermediate prognosis)
Drug: ABVD regimen — Given IV
  Arms: Group 1 (favorable prognosis); Group 2 (intermediate prognosis)
Drug: carmustine — Given IV
Drug: cisplatin — Given IV
  Arms: Group 3 (poor prognosis)
Drug: cytarabine — Given IV
  Arms: Group 3 (poor prognosis)
Drug: dacarbazine — Given IV
  Arms: Group 1 (favorable prognosis); Group 2 (intermediate prognosis)
Drug: dexamethasone — Given orally
  Arms: Group 3 (poor prognosis)
Drug: doxorubicin hydrochloride — Given IV
Drug: etoposide — Given IV
Drug: gemcitabine hydrochloride — Given IV
  Arms: Group 3 (poor prognosis)
Drug: ifosfamide — Given IV
  Arms: Group 3 (poor prognosis)
Drug: melphalan — Given IV
  Arms: Group 3 (poor prognosis)
Drug: methylprednisolone — Given IV
Drug: mitoguazone — Given IV
  Arms: Group 3 (poor prognosis)
Drug: vincristine sulfate — Given IV
  Arms: Group 1 (favorable prognosis); Group 2 (intermediate prognosis)
Drug: vindesine — Given IV
Drug: vinorelbine tartrate — Given IV
  Arms: Group 3 (poor prognosis)
Procedure: allogeneic hematopoietic stem cell transplantation — Patients undergo allogeneic stem cell transplantation
  Arms: Group 3 (poor prognosis)
Procedure: autologous hematopoietic stem cell transplantation — Patients undergo autologous stem cell transplantation
  Arms: Group 3 (poor prognosis)

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving drugs in different combinations may kill more cancer cells. It is not yet know which treatment regimen is more effective in treating Hodgkin lymphoma.

PURPOSE: This phase III trial is studying three different therapy regimens to compare how well they work in treating patients with previously untreated Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate event-free survival.

Secondary

* Evaluate overall survival.
* Evaluate the prognostic value of FDG-PET scanning.
* Evaluate progression-free survival.
* Evaluate tolerability.
* Evaluate rate of relapse.

OUTLINE: This is a multicenter study. Patients are assigned to 1 of 3 treatment groups according to prognosis.

* Group 1 (favorable prognosis): Patients receive ABVD chemotherapy comprising doxorubicin hydrochloride IV, bleomycin sulfate IV, vincristine sulfate IV, dacarbazine IV, and methylprednisolone IV on days 1 and 14. Treatment repeats every 28 days for 2 courses. Patients then undergo PET scan for evaluation of response. Patients receive additional treatment according to response.

  * Favorable response: Patients with favorable response receive 1 additional course of ABVD chemotherapy.
  * Unfavorable response: Patients with unfavorable response receive 1 course of VABEM chemotherapy comprising vindesine IV continuously on days 1-5, doxorubicin hydrochloride IV continuously on days 1-3, carmustine IV on day 3, etoposide IV on days 3-5, and methylprednisolone IV on days 1-5.
* Group 2 (intermediate prognosis): Patients receive 2 courses of ABVD chemotherapy. Patients then undergo PET scan for evaluation of response. Patients receive additional treatment according to response.

  * Favorable response: Patients with favorable response receive 4 additional courses of ABVD chemotherapy.
  * Unfavorable response: Patients with unfavorable response receive VABEM chemotherapy. Treatment with VABEM chemotherapy repeats every 28 days for 2 courses.
* Group 3 (poor prognosis): Patients receive 2 courses of VABEM chemotherapy. Patients then undergo PET scan for evaluation of response. Patients receive additional treatment according to response.

  * Favorable response: Patients with favorable response receive 1 additional course of VABEM chemotherapy.
  * Unfavorable response: Patients with unfavorable response receive CEO chemotherapy comprising cisplatin IV continuously on days 1-3, gemcitabine hydrochloride IV on days 1 and 8, and oral dexamethasone once daily on days 1-4. Treatment repeats every 21 days for 3 courses. Patients then undergo PET scan. Patients receive additional treatment according to response.

    * Favorable response: Patients with favorable response receive BEAM chemotherapy comprising carmustine IV on day -7, etoposide IV and cytarabine IV on days -6 to -3, and melphalan IV on day -2. Patients then undergo autologous stem cell transplantation on day 0.
    * Unfavorable response: Patients with unfavorable response receive MINE chemotherapy comprising mitoguazone IV, vinorelbine ditartrate IV, and ifosfamide IV on days 1-5 and etoposide IV on days 1-3. Treatment repeats every 28 days for 3 courses. Patients then undergo allogeneic or autologous stem cell transplantation.

Patients with favorable response or a "bulky" mass at diagnosis may also undergo radiotherapy.

After completion of study treatment, patients are followed periodically for 15 years.

ELIGIBILITY:
INCLUSION CRITERIA

* Life expectancy > 3 months
* LVEF normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Must be able to undergo follow-up for ≥ 15 years
* No impaired cardiac function that would preclude the administration of an anthracycline
* No other prior or concurrent malignancy, except for carcinoma in situ of the cervix or basal cell skin cancer
* No respiratory, kidney, or liver failure or other severe clinical insufficiency that would preclude study treatment
* No HIV or hepatitis B virus positivity
* No other disease that would preclude treatment with chemotherapy or radiotherapy

EXCLUSION CRITERIA:

* No concurrent participation in another experimental trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2008-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Event-free survival | treatments evaluation
  event free survival

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Senecal, Principal Investigator — French Innovative Leukemia Organization
Locations (1):
- FILO French Innovative Leukemia Organization, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided